CLINICAL TRIAL: NCT02252406
Title: Impact of Ranolazine on Inflammatory, Thrombogenic, Lipogenic, Biomarkers in Women With Angina and Metabolic Syndrome.
Brief Title: Impact of Ranolazine in Blood Markers in Women With Angina and Metabolic Syndrome
Acronym: IRMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WIRB20141202
Record Dates: First submitted 2014-08-11; First posted 2014-09-30 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Stable Angina; Metabolic Syndrome
Keywords: Stable Angina; Metabolic Syndrome; Women; Biomarkers
MeSH Terms: conditions — Angina, Stable; Metabolic Syndrome | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ranolazine (Experimental): Ranolazine would start with 500 mg BID and be force titrated to 1 gram po BID after 3 weeks. Down titration would only be allowed for side effects. This would be on top of all standard medical therapy.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo arm would start with 500 mg matching placebo tablet BID and be force titrated to 1 gram matching placebo tablet twice a day after 3 weeks. Down titration would only be allowed for side effects (if reported). This would be on top of all standard medical therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine 500 mg from baseline to week 3 and 1000 mg thereafter until week 24
  Other Names: Ranexa
  Arms: Ranolazine
Other: Placebo — Matching placebo tablets daily for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of ranolazine on different markers of cardiometabolic disease in women with stable angina.

DETAILED DESCRIPTION:
Evaluate the ability of ranolazine to favorably modify thrombogenic, inflammatory, lipogenic, oxidative stress and hormonal biomarkers in a relatively short period of time in a group of ethnically diverse women with chronic stable angina and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stable angina (> 3 months) on evidence based adequate therapy
* Evidence of stable coronary artery disease by any of these:
* MI, PCI or CABG > 30 days prior to enrollment or
* Angiography showing > 50% stenosis in major vessel, branch or bypass graft > 30 days of enrollment or
* Abnormal stress MPI nuclear study, or DBA stress echo where the decision has been to treat medically and where angina has remained stable for >= 3 months
* Evidence of the Metabolic Syndrome: As defined by ATP III criteria i.e 3/5 of following Abdominal circumference F > 88 cm (35 in), M > 102 cm (40 in) Hypertriglyceridemia ≥ 150 mg/dl HDL F < 50 mg/dl M < 40 mg/dl Blood Pressure ≥130/85 Fasting Glucose ≥100 mg/dl For reproductive age women, a negative urine pregnancy test is required if all other inclusion criteria are met.

Exclusion Criteria:

* Exclusion of patients with contraindications to use of RANEXA, including patients on CYP3A4 inducers/potent inhibitors, and patients with liver cirrhosis.
* Exclusion of Patients with CrCl < 30 mL/min
* Limit dose of RANEXA to 500mg BID in patients on concurrent diltiazem/ verapamil
* Limit concurrent simvastatin to 20 mg/day
* Limit concurrent metformin to 1700 mg/day Additional Exclusion
* Patients with variable -inconsistent symptoms
* Patients with unstable coronary artery disease or revascularization within 30 days of enrollment.
* Patients who have known severe liver disease.
* Patients already receiving maximal ranolazine therapy for more than 4 weeks
* Presence of diabetes (AIC≥ 6.5 and /or on insulin therapy or anti-diabetic medication other than metformin) unstable hypothyroidism, active infection, active cancer (or ongoing chemotherapy and/or radiation within a year who are not on remission) and/or recent major surgery or illness.
* Patients with any contraindication to ranolazine see above
* Women of reproductive age are excluded if they are planning to become pregnant in the next 6 -12 months after randomization.
* Patients who are pregnant or lactating
* Documented allergic reaction to ranolazine in the past.
* Unexplained prolongation of the QTc > 500 milliseconds.
* Current or planned co-administration of moderate CYP3A inhibitors (eg, diltiazem, verapamil, aprepitant, erythromycin, fluconazole, and grapefruit juice or grapefruit-containing products) is not a full contraindication, if meet inclusion criteria otherwise, these patients could be accepted in trial but dose will be limited to 500 mg BID as stated previously.
* Current or planned co-administration of strong CYP3A inhibitors (eg, ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir) OR strong CYP3A inducers (eg, rifampin, rifabutin, rifapentine, phenobarbital, phenytoin,carbamazepine, and St. John's Wort) is a contraindication.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12-17 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gladys P Velarde, MD, FACC, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 7/21/14 - 7/2/18 Location: UF Jacksonville Outpatient Cardiology clinic
Groups:
- Ranolazine: Ranolazine would start with 500 mg BID and be force titrated to 1 gram po BID after 3 weeks. Down titration would only be allowed for side effects. This would be on top of all standard medical therapy.
  Ranolazine: Ranolazine 500 mg from baseline to week 3
  Ranolazine: Ranolazine 1000mg daily at week 3 until weeks 24.
Period: Starting Dose Ranolazine 500 mg BID
Arm/Group | Ranolazine | Placebo
Started | 16 | 17
Completed | 12 | 14
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Titrated to Ranolazine 1000mg BID
Arm/Group | Ranolazine | Placebo
Started | 12 | 14
Completed | 9 | 13
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Impact of Ranolazine on Hemoglobin A1C
Description: Will evaluate the impact of ranolazine in HgbA1C in women with Metabolic Syndrome (MBS)
Time Frame: Change from baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Ranolazine Treated: We looked women randomized by table randomization to ranolazine that successfully titrated to maximum dose of tested drug (1,000 mg bid)
- Placebo: We looked women randomized by table randomization to placebo that successfully titrated to maximum dose of placebo drug
Arm/Group | Ranolazine Treated | Placebo
Number analyzed (Participants) | 9 | 13
percent change | -5 (6.2) | 2.6 (9.1)

2. Primary Outcome: Impact of Ranolazine on HDL-C Levels in Subjects
Description: Will evaluate the impact of ranolazine in HDL-C levels in women with metabolic syndrome
Time Frame: Change from Baseline to 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in HDL
Arm/Group | Ranolazine Treated | Placebo
Number analyzed (Participants) | 9 | 13
percentage of change in HDL | 6.6 (15.7) | 6.5 (46.6)

ADVERSE EVENTS:
Time Frame: Patients were followed for 24 weeks
Groups:
- Ranolazine Treated: Ranolazine would start with 500 mg BID and be force titrated to 1 gram po BID after 3 weeks. Down titration would only be allowed for side effects. This would be on top of all standard medical therapy
Arm/Group | Ranolazine Treated | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 3/16 | 0/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine Treated (N=16) | Placebo (N=17)
upset stomach (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02252406/Prot_SAP_000.pdf